CLINICAL TRIAL: NCT03559699
Title: An Open-Label Study To Evaluate the Efficacy and Safety of AG-348 in Regularly Transfused Adult Subjects With Pyruvate Kinase (PK) Deficiency
Brief Title: A Study Evaluating the Efficacy and Safety of AG-348 in Regularly Transfused Adult Participants With Pyruvate Kinase Deficiency (PKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG348-C-007; 2017-003803-22 (EudraCT Number)
Record Dates: First submitted 2018-03-26; First posted 2018-06-18 (Actual); Results first posted 2021-12-10 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Pyruvate Kinase Deficiency; Anemia, Hemolytic
MeSH Terms: conditions — Pyruvate Kinase Deficiency of Red Cells; Anemia, Hemolytic | interventions — mitapivat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AG-348 (Experimental): Participants received AG-348 tablets, administered orally, at a starting dose of 5 milligrams (mg), twice daily (BID), followed by two sequential dose level increases to 20 mg and 50 mg BID, for a period of 16 weeks in Part 1. This was followed by optimized dose BID, as determined by the investigator in Part 1, for a period of 24 weeks in Part 2.
  Interventions: Drug: AG-348

INTERVENTIONS:
Drug: AG-348 — Part 1 (Dose Optimization Period): Participants began by receiving 5 mg orally, BID. Each participant's dose of AG-348 was sequentially increased to 20 mg BID followed by 50 mg BID depending on their response to AG-348 and their tolerance.
  Part 2 (Fixed Dose Period): Optimized dose determined in Part 1.

SUMMARY:
Study AG348-C-007 was a multicenter study designed to evaluate the efficacy and safety of treatment with AG-348 in a minimum of 20, with up to 40, participants with pyruvate kinase (PK) deficiency, who were regularly receiving blood transfusions. The study was composed of two parts. During Part 1, Dose Optimization Period, participants started on a dose of 5 mg AG-348 administered twice daily. Over the course of Part 1 each participant's dose of AG-348 was sequentially increased to 20 mg twice a day, followed by 50 mg twice a day depending on their tolerance. During Part 2, Fixed-Dose Period, participants received AG-348 at their optimized dose from Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent;
* Male or female, aged 18 or older;
* Presence of at least 2 mutant alleles in the Pyruvate Kinase Liver and RBC (PKLR) gene, of which at least 1 is a missense mutation;
* History of a minimum of 6 transfusion episodes in the 52-week period prior to date of informed consent;
* Complete records of transfusion history for the 52 weeks prior to the date of informed consent, including all transfusion dates, number of blood units transfused for all the transfusions, and Hb concentrations within 1 week prior to transfusion for at least 80% of the transfusions;
* Have received at least 0.8 mg of oral folic acid daily for at least 21 days prior to the first dose of study drug, to be continued daily during study participation;
* Have adequate organ function;
* Negative serum pregnancy test for women of reproductive potential;
* For women of reproductive potential as well as fertile men and their partners who are women of reproductive potential: be abstinent or agree to use 2 forms of contraception, 1 of which must be considered highly effective, from the time of giving informed consent, during the study, and for 28 days following the last dose of AG-348;
* Willing to comply with all study procedures, in particular the individual transfusion trigger (TT) calculated based on 52 weeks of transfusion history, for the duration of the study.

Exclusion Criteria:

* Homozygous for the R479H mutation or have 2 non-missense mutations, without the presence of another missense mutation, in the PKLR gene;
* Significant medical condition that confers an unacceptable risk to participate in the study, and/or that could confound the interpretation of the study data;
* History of transfusions occurring on average more frequently than once every 3 weeks during the 52 weeks prior to date of informed consent;
* Splenectomy scheduled during the study treatment period or have undergone splenectomy within 12 months prior to signing informed consent;
* Currently enrolled in another therapeutic clinical trial. Prior participation in the PK Deficiency Natural History Study (NHS) (NCT02053480) or PK Deficiency Registry is permitted;
* Exposure to any investigational drug, device, or procedure within 3 months prior to the first dose of study drug;
* Prior bone marrow or stem cell transplant;
* Currently pregnant or breastfeeding;
* History of major surgery within 6 months of signing informed consent;
* Currently receiving medications that are strong inhibitors of CYP3A4, strong inducers of CYP3A4, strong inhibitors of P-glycoprotein (P-gp), or digoxin (a P-gp sensitive substrate medication) that have not been stopped for a duration of at least 5 days or 5 times their half-lives (whichever is longer) prior to start of study drug;
* Currently receiving hematopoietic stimulating agents (eg, erythropoietins [EPOs], granulocyte colony stimulating factors, thrombopoietins) that have not been stopped for a duration of at least 28 days prior to the first dose of study drug;
* History of allergy to sulfonamides if characterized by acute hemolytic anemia, drug induced liver injury, anaphylaxis, rash of erythema multiforme type or Stevens-Johnson syndrome, cholestatic hepatitis or other serious clinical manifestations;
* Allergy to AG-348 or its excipients;
* Currently receiving anabolic steroids, including testosterone preparations, within 28 days prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (19):
- United States (4):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Seattle Cancer Care Alliance, Seattle, Washington
- Toronto General Hospital, University Health Network, Toronto, Canada
- University of Copenhagen, Herlev Hospital, Herlev, Denmark
- France (2):
  - Hopital Universitaire Henri Mondor, Créteil
  - Hôpital de la Timone, Marseille
- St James's Hospital Department of Haematology, Dublin, Ireland
- Italy (4):
  - Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan
  - AORN Cardarelli, Napoli
  - Ospedale Galliera, Napoli
  - AOU Policlinico, Università della Campania "Luigi Vanvitelli", Napoli
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Department of Paediatrics and Thalassaemia Center, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand
- United Kingdom (4):
  - Addenbrooke's Hospital, Cambridge
  - Imperial College Healthcare NHS Trust, Hammersmith Hospital, London
  - University College London, London
  - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Samkari H, Grace RF, Glenthoj A, Andres O, Barcellini W, Galacteros F, Kuo KHM, Layton DM, Morado Arias M, Viprakasit V, Dong Y, Tai F, Hawkins P, Gheuens S, Morales-Arias J, Gilroy KS, Porter JB, van Beers EJ. Early-onset reduced bone mineral density in patients with pyruvate kinase deficiency. Am J Hematol. 2023 Mar;98(3):E57-E60. doi: 10.1002/ajh.26830. Epub 2023 Jan 9. No abstract available. PMID 36594181
- [Derived] Glenthoj A, van Beers EJ, Al-Samkari H, Viprakasit V, Kuo KHM, Galacteros F, Chonat S, Porter J, Zagadailov E, Xu R, Oluyadi A, Hawkins P, Gheuens S, Beynon V, Barcellini W; ACTIVATE-T investigators. Mitapivat in adult patients with pyruvate kinase deficiency receiving regular transfusions (ACTIVATE-T): a multicentre, open-label, single-arm, phase 3 trial. Lancet Haematol. 2022 Oct;9(10):e724-e732. doi: 10.1016/S2352-3026(22)00214-9. Epub 2022 Aug 18. PMID 35988546
- [Derived] Rab MAE, Van Oirschot BA, Kosinski PA, Hixon J, Johnson K, Chubukov V, Dang L, Pasterkamp G, Van Straaten S, Van Solinge WW, Van Beers EJ, Kung C, Van Wijk R. AG-348 (Mitapivat), an allosteric activator of red blood cell pyruvate kinase, increases enzymatic activity, protein stability, and ATP levels over a broad range of PKLR genotypes. Haematologica. 2021 Jan 1;106(1):238-249. doi: 10.3324/haematol.2019.238865. PMID 31974203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 27 participants were enrolled and treated in the study which was conducted across multiple sites in 9 countries: United States, Canada, Denmark, France, Ireland, Italy, Netherlands, Thailand, and United Kingdom. The study was conducted from 26 June 2018 to 12 November 2020.
Pre-assignment Details: Screening was done for a period of 8 weeks after the participant provided the informed consent. Investigators determined if the participants met all the inclusion criteria and none of the exclusion criteria to enroll in Part 1: Dose Optimization Period to receive AG-348 to determine the optimized dose followed by Part 2: Fixed Dose Period.
Period: Overall Study
Arm/Group | AG-348
Started | 27
Completed | 20
Not Completed | 7
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Groups:
- AG-348: Participants received AG-348 tablets, administered orally, at a starting dose of 5 mg, BID, followed by two sequential dose level increases to 20 mg and 50 mg BID, for a period of 16 weeks in Part 1. This was followed by optimized dose BID, as determined by the investigator in Part 1, for a period of 24 weeks in Part 2.
Arm/Group | AG-348
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (13.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Reduction in Transfusion Burden in Part 2
Description: Reduction in transfusion burden is defined as a ≥33% reduction in the number of RBC units transfused during the Fixed Dose Period standardized to 24 weeks compared with the historical transfusion burden standardized to 24 weeks (Standardized Control Period). The on-study (Fixed Dose Period) transfusion burden was calculated as the total number of transfused RBC units received in the Fixed Dose Period standardized to 24 weeks.
Time Frame: From Part 2, Day 1 to Part 2 Week 24
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AG-348
Number analyzed (Participants) | 27
percentage of participants | 37 [19.4 to 57.6]
Statistical Analysis 1: Comparison: AG-348; Test type: Other; p = 0.0002, Binomial exact test — 1-sided P-value

2. Secondary Outcome: Annualized Number of RBC Units Transfused During the Study
Description: The annualized total number of RBC units transfused during the entire study (both Part 1 and Part 2) is reported. It was calculated as the total number of RBC units transfused up to the end of Fixed Dose Period divided by the total number of days from the first dose date until the end date of Fixed Dose Period × 52.
Time Frame: Part 1 Day 1 to Part 2 Week 24
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: RBC units
Arm/Group | AG-348
Number analyzed (Participants) | 27
RBC units | 11.52 (10.543)

3. Secondary Outcome: Number of Transfusion Episodes in Part 2
Description: This is the number of transfusion episodes in Part 2. The number of transfusion episodes were standardized to 24 weeks. Transfusions received over up to 3 consecutive days were counted as 1 episode.
Time Frame: From Part 2 Day 1 to Part 2 Week 24
Population: Full analysis set included all participants who received at least 1 dose of study drug. Number analyzed is the number of participants evaluated for the outcome measure.
Measure: Mean (Standard Deviation); unit: transfusion episodes
Arm/Group | AG-348
Number analyzed (Participants) | 26
transfusion episodes | 2.88 (2.694)

4. Secondary Outcome: Percentage of Transfusion-Free Participants in Part 2
Description: Transfusion-free responders were the participants who were transfusion-free in Part 2.
Time Frame: From Part 2 Day 1 to Part 2 Week 24
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AG-348
Number analyzed (Participants) | 27
percentage of participants | 22.2 [8.6 to 42.3]

5. Secondary Outcome: Percentage of Participants Achieving Normal Hemoglobin (Hb) Concentrations in Part 2
Description: This is the percentage of participants who achieved hemoglobin (Hb) concentrations in the normal range at least once, 8 weeks or more after a transfusion in Part 2.
Time Frame: From Part 2 Day 1 to Part 2 Week 24
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AG-348
Number analyzed (Participants) | 27
percentage of participants | 11.1 [2.4 to 29.2]

6. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the study drug. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Through 4 weeks after last dose (approximately Part 2, Week 31)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | AG-348
Number analyzed (Participants) | 27
percentage of participants | 100

7. Other Pre Specified Outcome: Percentage of Participants Experiencing an Adverse Event of Special Interest (AESI)
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AESI can be serious or non-serious.
Time Frame: From Part 1 Day 1 to end of Part 2, including follow-up (Day 197)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Bone Mineral Density Z-Score
Time Frame: Part 1, Day 1, Part 2, Day 1 and Part 2, Week 24
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Bone Mineral Density T-Score
Time Frame: Part 1, Day 1, Part 2, Day 1 and Part 2, Week 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From Part 1 Day 1 to end of Part 2, including follow-up (up to Day 197)
Description: Safety analysis set included all participants who received at least 1 dose of the study drug.
Arm/Group | AG-348
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 3/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AG-348 (N=27)
Blood Triglyceride Increased (Investigations) | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1
Renal Colic (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AG-348 (N=27)
Nasopharyngitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Viral upper respiratory tract infection (Infections and infestations) | 4
Influenza (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Suspected COVID-19 (Infections and infestations) | 2
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Alanine aminotransferase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 5
Liver iron concentration increased (Investigations) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Fatigue (General disorders) | 5
Initial insomnia (Psychiatric disorders) | 2
Middle insomnia (Psychiatric disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Vaginal haemorrhage (Reproductive system and breast disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The information obtained from the clinical study will be used towards the development of AG-348 and may be disclosed to regulatory authority(ies), other Investigators, corporate partners, or consultants as required.

DOCUMENTS (2):
  • Study Protocol (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT03559699/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT03559699/SAP_001.pdf